CLINICAL TRIAL: NCT01330992
Title: Human Circadian Sensitivity to Very Short Light Pulses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth B. Klerman, Associate Professor, Associate Physician, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NIH-RC2-HL101340
Record Dates: First submitted 2011-04-01; First posted 2011-04-07 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Circadian Rhythm Disorders
Keywords: Circadian rhythms; Melatonin; Ocular light exposure; Darkness Exposure; Performance; Alertness
MeSH Terms: conditions — Chronobiology Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ocular Light or Dark Exposure (Experimental): Ocular Light or Dark Exposure
  Interventions: Other: Ocular light or darkness exposure

INTERVENTIONS:
Other: Ocular light or darkness exposure — Ocular light or darkness exposure

SUMMARY:
The mammalian eye serves both visual and non-image-forming functions. New information about the non-image-forming anatomy and physiology of the eye has revealed effects of ocular light stimuli on human circadian rhythms, melatonin suppression, heart rate, pupillary reflexes, cognitive performance, alertness and sleep. The results of the proposed work can be used to make predictions about the effects of light, to make recommendations involving exposure to or avoidance of light, and to design environmental lighting, resulting in improved health and alertness and decreased errors and accidents.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* No medications
* No eye disease
* No sleep disorders
* No psychiatric disorders

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Circadian Phase (hours) | Before and after intervention (day 1)
  Circadian phase (hours) measured before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States